CLINICAL TRIAL: NCT00097383
Title: A Phase 2 Study of Alimta and Epirubicin Administered Every 21 Days in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Study of Alimta and Epirubicin Administered in Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 4028; H3E-MC-JMDU
Record Dates: First submitted 2004-11-22; First posted 2004-11-23 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Epirubicin

INTERVENTIONS:
Drug: ALIMTA plus Epirubicin

SUMMARY:
This is a non-randomized Phase 2 portion of a study testing ALIMTA and epirubicin in combination for locally advanced or metastatic breast cancer. Epirubicin is a well-established drug for the therapy of breast cancer. Both ALIMTA and epirubicin have been combined with other drugs but they have not yet been combined with each other. It is expected that the patient will benefit from the different mechanisms of action of the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic breast cancer not amenable to local treatment.
* Patients must be chemo-naive or have only neoadjuvant and/or adjuvant chemotherapy.
* Patients must have at least one measurable lesion in an area not previously irradiated.
* No chemotherapy at least 4 weeks prior to study enrollment.
* Signed informed consent from patient.

Exclusion Criteria:

* Treatment with any drug within the last 30 days that has not received regulatory approval.
* Serious systemic disorders, including active infection.
* Significant cardiovascular disease.
* Pregnancy or breast feeding.
* Inability or unwillingness to take folic acid or Vitamin B12 supplementation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (25):
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., La Plata, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Rosario, Santa Fe Province
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ciudad de Buenos Aires
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Wilrijk
- Brazil (7):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Maceió, Alagoas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Belo Horizonte, BH
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Curitiba, Paraná
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Porto Alegre, Rio Grande do Sul
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., São Paulo, Sao Paulo/SP
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., São Paulo, São Paulo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sorocaba, São Paulo
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Guadalajara, Jalisco
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mexico City, Mexico City
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Col. Campestre Churubusco
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mexico City
- Portugal (7):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Arquiparque-Miraflores, Alges
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Porto
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Proto
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Santa Maria da Feira
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Santarém